CLINICAL TRIAL: NCT04832282
Title: Feasibility of a New Method Named Napoleon to Measure Gastrojejunal Anastomosis in Gastric Bypass Patients With Weight Regain
Brief Title: Napoleon Measurement of Gastrojejunal Anastomosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20-01436
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Gastric Bypass; Weight Regain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Roux-en-Y gastric bypass patients with weight regain (Other): The study population is Roux-en-Y gastric bypass (RYGB) patients with weight regain undergoing an endoscopy at Bellevue Hospital Center or Brigham and Women's Hospital.
  Interventions: Device: Napoleon; Other: Visual estimation

INTERVENTIONS:
Device: Napoleon — The Micro-Tech Endoscopic Measurement Device named Napoleon is a small catheter with a 30mm ruler calibrated at 1mm intervals with 5mm demarcations. It is classified as a Class 1, 510(k) exempt device by the FDA. The device was originally intended to measure polyps. However, it is used off-label in this study and is considered investigational.
Other: Visual estimation — For each case, endoscopists will first visually estimate the diameter of the GJA by comparing its size to the upper endoscope.

SUMMARY:
This is a clinical trial assessing the feasibility of the Napoleon device for measuring the gastrojejunal anastomosis (GJA). The study population is Roux-en-Y gastric bypass (RYGB) patients with weight regain undergoing an endoscopy at Bellevue Hospital Center or Brigham and Women's Hospital. investigators aim for a sample size of up to 100 cases. For each case, endoscopists will first visually estimate the diameter of the GJA by comparing its size to the upper endoscope. Then, they will measure the GJA with Napoleon. Investigators will compare the GJA measurements performed using visual estimation and Napoleon. A survey will be given to all endoscopists to assess the level of ease using Napoleon.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. RYGB patient with weight regain age 18-90
2. Scheduled for an endoscopy
3. Willingness and ability to provide informed consent

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. History of prior endoscopies with complications

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean difference in measured Gastrojejunal Anastomosis size between Napoleon and visual estimation | 8 months

SECONDARY OUTCOMES:
Proportion of cases with different recommended endoscopic treatment based on GJA size measured by Napoleon Device | 8 months
Level of ease with using Napoleon in terms of placement, extension/retraction, and photo acquisition | 8 months
Additional procedure time needed to incorporate use of Napoleon | 8 months
Proportion of cases with adverse events or unanticipated problems related to use of Napoleon | 8 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Bellevue Hospital Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Violeta.Popov@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements
Access Criteria: Requests may be directed to: Violeta.Popov@nyulangone.org.